CLINICAL TRIAL: NCT05531773
Title: Assessment of Post COVID-19 Manifestations in a Multicenter Cohort Study (EuCARE-POSTCOVID Study)
Brief Title: Post COVID-19 Condition
Status: Recruiting | Type: Observational
Sponsor: Euresist Network GEIE (Other)
Collaborators: ASST Santi Paolo e Carlo (Other); Vilnius University Hospital Santaros Klinikos (Other); Heinrich-Heine University, Duesseldorf (Other); University of Rome Tor Vergata (Other); Hospital Regional de Alta Especialidad "Dr. Juan Graham Casasus" (Other); St Mary's Hospital, London (Other); Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Sponsor
Other Study IDs: EuCARE - PostCOVID
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples and a nasopharyngeal swab at COVID-19 diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 patients: patients recovered from an acute COVID-19 episode
  Interventions: Other: follow up of COVID-19 Patients

INTERVENTIONS:
Other: follow up of COVID-19 Patients — In each participating center a post COVID-19 outpatient clinic is already working or will be settled up to care COVID-19 patients after the acute phase. At the post COVID-19 clinic patients will undergo routine blood exams and will be visited by Infectious Diseases physicians after recovery from the acute episode of COVID-19 disease. According to the clinical issues of the patients and the procedures of the study, if necessary, the patients will be visited by other practitioners (Pneumologists, Cardiologists, Neurologists, Physiatrist and Psychologists or others).
  Patients who have been already visited at the post COVID outpatient clinics from 01/03/2020 and for whom data of the acute phase and the follow up have been collected will be enrolled in the study and retrospectively analyzed.

SUMMARY:
The EuCARE-POSTCOVID study is an observational multicentre study enrolling COVID-19 patients recovered from the acute phase of disease to investigate the prevalence and possible predictors of post COVID-19 condition. The study will retrospectively analyze data already collected at the post COVID-19 outpatients services of the participating centers; furthermore, a prospective cohort study will be performed.

DETAILED DESCRIPTION:
Background:

The EuCARE project includes several cohorts of patients and schools to provide an advance response to COVID-19 epidemics. The cohorts belong to different geographic areas including European countries, Kenya, Mexico, Russia and Vietnam, and will consolidate or expand interactions with other cohorts. A comprehensive multidisciplinary team of clinicians, virologists, epidemiologists, statisticians and top experts in artificial intelligence will collaborate to investigate:

* the natural and artificial immunity to the different viral variants in health care workers;
* the clinical course and long-term follow up of hospitalized COVID-19 patients to derive the role of different viral variants in the outcome of the infection, including post COVID-19 condition;
* the best strategies to control the spread of different viral variants in schools, by comparing the outcome of diverse containment and prevention measures in relation to the prevalence and dynamics of the variants.

Post COVID-19 condition is defined as the persistence or new onset of symptoms 3 months after an acute episode of COVID-19; these symptoms could last 2 or even more months and are not explained by an alternative diagnosis. The prevalence of these ongoing symptoms is very variable among the different studies, but seems high, affecting up to 50-60% of recovered patients.

Moreover, the post COVID-19 condition is described more commonly in females and more severe patients, but can be observed at all ages and in patients with a mild acute episode of COVID-19 disease.

AIMS AND OBJECTIVES The hypothesis of the study is that a relatively high proportion of patients recovered from an acute COVID-19 episode develops long-term sequelae, defined as the presence of ongoing or new onset physical and/or psychological symptoms at three months after the acute illness. These symptoms could last at least two months or even longer.

The mechanisms underpinning the post-acute and chronic manifestations of COVID-19 are not entirely understood.

The predictors of post COVID-19 condition have not yet identified, but the first evidence suggest that patients experiencing persistent symptoms, at 4-weeks or 8-weeks after the acute disease, were more likely elderly, females and hospitalized in the acute phase compared to the patients reporting symptoms for a short period of time (Carole et al, 2021).

We also hypothesized that older age, female gender, severity of disease and previous patients' comorbidities could be risk factors for the development of post COVID-19 condition.

Finally, our hypothesis is that the new variant "Omicron" could be associated with a lower inflammation and disease's severity during the acute phase and, thus, with a lower incidence of post COVID-19 condition.

Study objective:

Primary objective is to assess the incidence and risk factors of post COVID-19 condition in a cohort of recovered COVID-19 patients.

Secondary objectives are:

to evaluate the association between circulating SARS-CoV-2 variants and risk of post COVID-19 condition; to evaluate long-term residual organ damage (lung, hearth, Central Nervous System, CNS, Peripheral Nervous System, PNS) in relation to patient's characteristics and virology (variant, viral load in the acute phase).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >18 years old;
* Confirmed diagnosis of COVID-19 disease (positive SARS CoV-2 RNA on naso- pharyngeal swab or upper respiratory sample);
* Mild COVID-19 disease without hospital admission or moderate/severe disease requiring hospital admission for COVID-19 or hospitalization for other medical issues with a positive SARS CoV-2 RNA sample;
* Informed consent for the study.

Exclusion Criteria:

* death during hospitalization:
* patient's decline to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute COVID-19 disease from 01/03/2020 to 01/02/2025 at the participating centers will be enrolled in the study; two groups of patients recovered from acute COVID-19 will be enrolled:
  * Group 1 (hospitalized patients): patients hospitalized for COVID-19 disease;
  * Group 2 (outpatients): patients diagnosed with mild COVID-19 disease and thus not hospitalized (these patients will be referred to the Clinic of Infectious Diseases by the general practitioner or have received monoclonal antibodies for COVID-19 or antiviral treatments for COVID-19 at the Clinic of Infectious Diseases or have been visited at the Emergency Department of the hospital).
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of post COVID-19 condition | through study completion, an average of 3 years
Persistence of post COVID-19 condition beyond 2-3 months from the acute COVID-19 disease | through study completion, an average of 3 years
Predictors of post COVID-19 condition | through study completion, an average of 3 years
Long-term organ damage (lung, heart, Central Nervous System, Peripheral Nervous System) associated with post COVID-19 condition | through study completion, an average of 3 years
Virological and immunological phenotype of post COVID-19 condition | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: ANTONELLA D'ARMINIO MONFORTE, PROF, Study Chair — ASST SANTI GIOVANNI E CARLO
Locations (7):
- University Hospital Heinrich Heine, Düsseldorf, Germany
- Italy (2):
  - Policlinico "Tor Vergata", Università degli Studi di Roma TOR VERGATA, Rome, Lazio
  - ASST Santi Paolo e Carlo, Milan, Lombardy
- Vilnius University Hospital, Santaros Klinikos, Vilnius, Lithuania
- Regional Hospital Dr. Juan Graham Casasús, Villahermosa, Tabasco, Mexico
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal
- St. Mary Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study is part of a project funded by the European Commission and the project agreement with theCommission affirms that the data and the results will be public
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: AFTER THE STUDY END NO TIME LIMIT WAS FIXED
Access Criteria: REQUEST TO THE STUDY COORDINATOR OR TO THE PROJECTPARTNERS
URL: https://eucareresearch.eu/

REFERENCES:
- [Derived] Varisco B, Bai F, De Benedittis S, Tavelli A, Cozzi-Lepri A, Sala M, Miraglia FG, Santoro MM, Ceccherini-Silberstein F, Shimoni Y, Ravid S, Kozlovski T, Konig F, Pfeifer N, Shamsara E, Parczewski M, Monforte AD, Incardona F, Mommo C, Marchetti G. EuCARE-POSTCOVID Study: a multicentre cohort study on long-term post-COVID-19 manifestations. BMC Infect Dis. 2023 Oct 13;23(1):684. doi: 10.1186/s12879-023-08595-0. PMID 37833640